CLINICAL TRIAL: NCT02380027
Title: A Randomized Control Trial of Magnetic Resonance Imaging-targeted Biopsy Compared to Standard Trans-rectal Ultrasound Guided Biopsy for the Diagnosis of Prostate Cancer in Men Without Prior Biopsy
Brief Title: PRostate Evaluation for Clinically Important Disease: Sampling Using Image-guidance Or Not?
Acronym: PRECISION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University Hospital, Lille (Other); Radboud University Medical Center (Other); London North West Healthcare NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Sunnybrook Health Sciences Centre (Other); University College London Hospitals (Other); University Ghent (Other); Helsinki University Central Hospital (Other); Jewish General Hospital (Other); University of Roma La Sapienza (Other); Göteborg University (Other); Erasmus Medical Center (Other); Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency); University Hospital Heidelberg (Other); University Hospital, Aachen (Other); Hampshire Hospitals NHS Foundation Trust (Other); Princess Alexandra Hospital NHS Trust (Other); San Raffaele University Hospital, Italy (Other); M.D. Anderson Cancer Center (Other); University Hospital Southampton NHS Foundation Trust (Other); University of Oulu (Other); The Whittington Hospital NHS Trust (Other Government); University Hospital of Cologne (Other); Mayo Clinic (Other); Centro de Urologia Argentina (Unknown); Weill Medical College of Cornell University (Other); University of Chicago (Other); University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Veeru Kasivisvanathan, Study Coordinator, University College, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DRF-2014-07-146
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Prostate Neoplasm
Keywords: Prostate biopsy; MRI; transrectal; Detection
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI-arm (Experimental): Men in this arm will undergo multi-parametric MRI. In the presence of a suspicious area, a man will undergo MRI-targeted biopsy with cores targeted to the suspicious lesion. In the absence of a suspicious area, no biopsy will be taken.
  Interventions: Device: MRI; Procedure: MRI-targeted biopsy
- TRUS-biopsy arm (Active Comparator): Men in this arm undergo standard 12-core trans-rectal ultrasound guided prostate biopsy
  Interventions: Procedure: TRUS-biopsy

INTERVENTIONS:
Device: MRI — This will be a multi-parametric MRI of the prostate
  Arms: MRI-arm
Procedure: MRI-targeted biopsy — This will be a biopsy targeted to suspicious areas on the MRI
  Arms: MRI-arm
Procedure: TRUS-biopsy — This will be a standard 12 core trans-rectal prostate biopsy
  Arms: TRUS-biopsy arm

SUMMARY:
This evaluates the detection rates of prostate cancer by MRI-targeted prostate biopsy compared to standard 12-core trans-rectal ultrasound guided (TRUS) prostate biopsy. Each participant will be randomly allocated to one of the biopsy tests.

We hypothesise that MRI-targeted biopsy will detect no fewer clinically significant cancers than TRUS biopsy but will detect fewer clinically insignificant prostate cancers than TRUS biopsy.

DETAILED DESCRIPTION:
The classical pathway for the diagnosis of prostate cancer is trans-rectal ultrasound guided (TRUS) biopsy of the prostate following a raised PSA. This is currently the mainstay for prostate cancer diagnosis in the majority of centres. It has many advantages and can be performed routinely under local anaesthetic in an outpatient setting. However it does have some limitations, including the over-diagnosis of insignificant cancer and the under-diagnosis of significant cancer.

An alternative pathway for the diagnosis of prostate cancer in men with raised prostate specific antigen (PSA) is to perform a multi-parametric MRI to localize cancer and to use this information to influence conduct of a subsequent biopsy, known as an MRI-targeted biopsy. MRI-targeted biopsy has been shown in preliminary studies to detect a similar amount of clinically significant cancer to TRUS-biopsy but may have several advantages, for example in reducing the number of men who require biopsy.

This randomized controlled trial aims to assess the detection rate of clinically significant and clinically insignificant cancer of MRI-targeted biopsy compared to standard 12-core TRUS biopsy in men referred with clinical suspicion of prostate cancer who have had no prior prostate biopsy.

A 'clinically insignificant cancer' is cancer which is unlikely to progress or affect a man's life expectancy and therefore does not warrant treatment. However when diagnosed with insignificant cancer a large proportion of patients request treatment in case a more significant cancer is present. A prostate cancer detection pathway that finds significant cancers while avoiding the diagnosis of insignificant cancer is a major unmet need.

The potential implications of this trial include:

* A redefining of the prostate cancer diagnostic pathway
* A reduction in the number of patients undergoing prostate biopsy
* A reduction in the number of biopsy cores taken per patient
* A reduction in biopsy-related sepsis, pain and other side effects
* A reduction in the over-diagnosis of clinically insignificant prostate cancer
* A reduction of the economic burden of diagnosing and treating prostate cancer

ELIGIBILITY:
Inclusion Criteria:

1. Men at least 18 years of age referred with clinical suspicion of prostate cancer who have been advised to have a prostate biopsy
2. Serum PSA ≤ 20ng/ml within the previous 3 months
3. Suspected stage ≤ T2 on rectal examination (organ-confined prostate cancer) within the previous 3 months
4. Fit to undergo all procedures listed in protocol
5. Able to provide written informed consent

Exclusion Criteria:

1. Prior prostate biopsy
2. Prior treatment for prostate cancer
3. Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated glomerular filtration rate ≤ 50mls/min)
4. Contraindication to prostate biopsy
5. Men in whom artifact would reduce the quality of the MRI
6. Previous hip replacement surgery, metallic hip replacement or extensive pelvic orthopaedic metal work
7. Unfit to undergo any procedures listed in protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of men with clinically significant detected | When histology results available, at an expected average of 30 days post-biopsy

SECONDARY OUTCOMES:
Proportion of men in MRI arm who avoid biopsy | When MRI results available, at an expected average of 30 days post-MRI
Proportion of men with MRI score 3, 4 or 5 who have no clinically significant cancer detected | When histology results available, at an expected average of 30 days post-biopsy
Proportion of men who go on to definitive treatment for prostate cancer | After treatment decision, at an expected average of 30 days post-biopsy
  Definitive treatment can be localised (e.g. radical prostatectomy, radiotherapy, brachytherapy) or systemic (hormone therapy, chemotherapy)
Cancer core length of the most involved biopsy core (maximum cancer core length) | When histology results available, at an expected average of 30 days post-biopsy
  Cancer core length in mm
Proportion of men with post-biopsy adverse events | 30 days post biopsy
EQ-5D-5L Quality of Life scores | Baseline, 24 hours post intervention and 30 days post intervention
  EQ-5D gives a measure of health-related quality of life. The descriptive system gives a weighted index score from 0-1 where 1 is perfect health and 0 is the worst health possible. The visual analogue score is a measure of overall self-rated health status where 100 is the best imaginable health state and 0 is the worst imaginable health state.
Proportion of men undergoing Radical prostatectomy who have Gleason grade upgrading | An expected average of 90 days post-biopsy
Cost per diagnosis of cancer | 30 days post-biopy
Proportion of men with clinically insignificant detected | When histology results available, at an expected average of 30 days post-biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Moore, MD FRCS, Study Chair — University College Hospital London and University College London; Mark Emberton, MD FRCS, Study Chair — University College Hospital London and University College London
Locations (1):
- University College Hospitals, London, United Kingdom

REFERENCES:
- [Derived] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Derived] Kasivisvanathan V, Jichi F, Klotz L, Villers A, Taneja SS, Punwani S, Freeman A, Emberton M, Moore CM. A multicentre randomised controlled trial assessing whether MRI-targeted biopsy is non-inferior to standard transrectal ultrasound guided biopsy for the diagnosis of clinically significant prostate cancer in men without prior biopsy: a study protocol. BMJ Open. 2017 Oct 12;7(10):e017863. doi: 10.1136/bmjopen-2017-017863. PMID 29025845